CLINICAL TRIAL: NCT00335049
Title: Study of Theories About Myopia Progression (STAMP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Karla Zadnik, OD PhD / Principal Investigator, The Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2005H0157; K12EY015447 (NIH)
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Myopia
Keywords: myopia progression; bifocal
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAL (Experimental): Progressive Addition Spectacle Lenses (PALs) with a +2.00 D add worn for first year off study. Single Vision Lenses worn for second year of study.
  Interventions: Device: progressive addition spectacle lens (bifocal)
- SVL (Active Comparator): Single Vision Lenses (SVLs) worn both years of the study.
  Interventions: Device: Single Vision Lenses (SVLs)

INTERVENTIONS:
Device: progressive addition spectacle lens (bifocal) — Progressive addition lenses (PAL) with a +2.00 D add.
  Other Names: PAL
  Arms: PAL
Device: Single Vision Lenses (SVLs) — Single vision spectacle lenses.
  Other Names: SVL
  Arms: SVL

SUMMARY:
At this time, we do not know what causes a child to become more nearsighted (myopic). STAMP will help us better understand nearsightedness in children. Children will be randomly chosen to wear regular glasses (single vision lenses) or no-line bifocal glasses (progressive addition lenses) for the first year of the study. All children will wear regular glasses for the second year of the study. STAMP will compare how the eye changes shape in the two groups to help us understand why children become nearsighted. The two theories of myopia progression that are being evaluated are based on different factors. One theory is based on environmental factors such as extended near work while the other theory is based on genetically coded factors.

DETAILED DESCRIPTION:
Eligible children will be enrolled, randomized, and followed at six-month intervals for two years with all children wearing single vision lenses for the second year. At each visit, complete measurements of the components of the eye will be made to explain the mechanism responsible for the Progressive Addition Lens (PAL) treatment effect and why it occurs mainly during the first year of bifocal wear (Gwiazda et al. 2003). While hyperopic retinal blur (blur at the back of the eye) due to accommodative lag (poor focusing when doing close work) has been proposed as a possible mechanism driving myopia progression (Gwiazda et al. 1993), others have shown that accommodative lag accompanies rather than precedes the onset of myopia (Mutti et al., 2006). This suggests that accommodative lag is a result of another possible mechanism resulting in myopia progression such as crystalline lens-induced ciliary-choroidal tension (a model in which the lens in the eye is stretched and is not as good at focusing up close) (Mutti et al., 2000). According to this proposed mechanism, high accommodative lag in myopia results from increased crystalline lens tension that is transmitted through the choroid (an outside layer of the eye). This tension results in restricted equatorial (the vertical dimension of the eye) eye growth with no axial (front to back) restriction to eye growth and yields a prolate ocular shape (an eye that is longer than it is wide) in myopes (Mutti et al., 2000).

Comparisons: Refractive error (glasses prescription), axial length (length of the eye), peripheral eye shape, accommodation (focusing ability), corneal shape (shape of the front of the eye), anterior chamber depth, crystalline lens thickness and curvatures (shape of the lens in the eye), central and peripheral higher-order aberrations (how well light focuses in the eye), and phoria (eye alignment) will be measured at six-month intervals. The primary study outcome is refractive error measured by cycloplegic autorefraction. Comparison of the biometric data collected both during the first year when the PAL intervention is present and during the second year when the PAL intervention is removed will allow us to differentiate between the two theories under consideration. We will also evaluate whether the modest PAL treatment effect that has been reported during the first year of PAL wear is permanent.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 11 years of age
* Best corrected vision of at least 20/30 in each eye
* Birth weight > 1250g

(The criteria below will be evaluated at a screening visit to find out if the child can participate)

* Accommodative lag >= 1.30 D (for a 4D stimulus)
* At least -0.75 D myopia in each meridian measured with cycloplegic autorefraction but not more than -4.50 D in each meridian in each eye
* Esophoria at near if more than -2.25 D spherical equivalent (high myopia)
* Astigmatism < 2.00 DC in each eye
* Anisometropia < 2.00 D

Exclusion Criteria:

* Strabismus (eye turn)
* History of contact lens wear
* History of previous bifocal wear
* Diabetes mellitus

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2006-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Cycloplegic autorefraction | Baseline, 6, 12, 18, and 24 months

SECONDARY OUTCOMES:
Phoria | Baseline, 6, 12, 18, and 24 months
Accommodative lag | Baseline, 6, 12, 18, and 24 months
AC/A ratio | Baseline, 6, 12, 18, and 24 months
Corneal shape and thickness | Baseline, 6, 12, 18, and 24 months
Intraocular pressure | Baseline, 6, 12, 18, and 24 months
Peripheral ocular shape | Baseline, 6, 12, 18, and 24 months
Central and peripheral aberrations | Baseline, 6, 12, 18, and 24 months
Crystalline lens thickness and curvature | Baseline, 6, 12, 18, and 24 months
Anterior chamber depth | Baseline, 6, 12, 18, and 24 months
Axial length | Baseline, 6, 12, 18, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: David A Berntsen, OD, PhD, Principal Investigator — University of Houston; Karla Zadnik, OD, PhD, Principal Investigator — Ohio State University; Donald O Mutti, OD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States

REFERENCES:
- [Background] Gwiazda J, Thorn F, Bauer J, Held R. Myopic children show insufficient accommodative response to blur. Invest Ophthalmol Vis Sci. 1993 Mar;34(3):690-4. PMID 8449687
- [Background] Gwiazda J, Hyman L, Hussein M, Everett D, Norton TT, Kurtz D, Leske MC, Manny R, Marsh-Tootle W, Scheiman M. A randomized clinical trial of progressive addition lenses versus single vision lenses on the progression of myopia in children. Invest Ophthalmol Vis Sci. 2003 Apr;44(4):1492-500. doi: 10.1167/iovs.02-0816. PMID 12657584
- [Background] Mutti DO, Sholtz RI, Friedman NE, Zadnik K. Peripheral refraction and ocular shape in children. Invest Ophthalmol Vis Sci. 2000 Apr;41(5):1022-30. PMID 10752937
- [Background] Mutti DO, Mitchell GL, Hayes JR, Jones LA, Moeschberger ML, Cotter SA, Kleinstein RN, Manny RE, Twelker JD, Zadnik K; CLEERE Study Group. Accommodative lag before and after the onset of myopia. Invest Ophthalmol Vis Sci. 2006 Mar;47(3):837-46. doi: 10.1167/iovs.05-0888. PMID 16505015
- [Derived] Lawrenson JG, Shah R, Huntjens B, Downie LE, Virgili G, Dhakal R, Verkicharla PK, Li D, Mavi S, Kernohan A, Li T, Walline JJ. Interventions for myopia control in children: a living systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 16;2(2):CD014758. doi: 10.1002/14651858.CD014758.pub2. PMID 36809645
- [Derived] Berntsen DA, Barr CD, Mutti DO, Zadnik K. Peripheral defocus and myopia progression in myopic children randomly assigned to wear single vision and progressive addition lenses. Invest Ophthalmol Vis Sci. 2013 Aug 27;54(8):5761-70. doi: 10.1167/iovs.13-11904. PMID 23838771
- [Derived] Berntsen DA, Sinnott LT, Mutti DO, Zadnik K. A randomized trial using progressive addition lenses to evaluate theories of myopia progression in children with a high lag of accommodation. Invest Ophthalmol Vis Sci. 2012 Feb 13;53(2):640-9. doi: 10.1167/iovs.11-7769. Print 2012 Feb. PMID 22205604
- [Derived] Berntsen DA, Mutti DO, Zadnik K. The effect of bifocal add on accommodative lag in myopic children with high accommodative lag. Invest Ophthalmol Vis Sci. 2010 Dec;51(12):6104-10. doi: 10.1167/iovs.09-4417. Epub 2010 Aug 4. PMID 20688729